CLINICAL TRIAL: NCT02298621
Title: The Effect of Pomegranate Juice Intake on Cardiometabolic Factors in Subjects With Metabolic Syndrome.
Brief Title: Pomegranate Juice and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Urmia University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1175
Record Dates: First submitted 2014-11-05; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2012-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pomegranate juice (Experimental): pomegranate juice: 500 ml
  Interventions: Other: pomegranate juice; Other: placebo
- placebo (Placebo Comparator): sugar + aroma+ color: 500ml
  Interventions: Other: pomegranate juice; Other: placebo

INTERVENTIONS:
Other: pomegranate juice — Randomized clinical trial or RCT
Other: placebo — Randomized clinical trial or RCT

SUMMARY:
The effect of pomegranate juice (PJ) intake on cardiovascular risks in subject with metabolic syndrome.

DETAILED DESCRIPTION:
The effect of pomegranate juice (PJ) intake on cardiovascular risks in subject with metabolic syndrome in shabestar.

ELIGIBILITY:
Inclusion Criteria:

* presence of ≥3 of the following diagnostic of MetS:

  * serum TGs of at least 150 mg/dL,
  * waist circumference of more than 102 cm (40 in) in men and more than 88 cm (35 in) in women,
  * high-density lipoprotein (HDL) level less than 40 mg/dL in men and less than 50 mg/dL in women,
  * blood pressure 135/85 mm Hg or higher, or
  * fasting glucose 100 mg/dL or Higher

Exclusion Criteria:

* liver cirrhosis,
* chronic pancreatitis,
* gastrointestinal or connective diseases,
* kidney stones, or
* renal failure,
* alcohol Consumption,
* having an allergy to pomegranate juice,
* a change in diet,
* the large increase in LDL so that required drug treatment.
* use of statins of fibrates, corticosteroids, nitrates, acetyl-salicylic acid or other anti-platelet drugs, oral hypoglycemic drugs, nonsteroidal anti-inflammatory drugs, or drugs interfering with coagulation;
* pregnancy or lactation in the past 6 mo, supplementation with vitamins or antioxidants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in values of metabolic syndrome components at 1 week | 1 week

SECONDARY OUTCOMES:
Change from baseline in values of insulin resistance (HOMA-IR), total cholesterol, LDL-C, VLDL-C and hs-CRP at 1 week | 1 weeks
  Insulin resistance via HOMA-IR

CONTACTS AND LOCATIONS:
Overall Officials: mohammad alizadeh, Study Director — Urmia University of Medical Sciences
Locations (1):
- Urmia University of Medical Sciences, Urmia, Iran